CLINICAL TRIAL: NCT05528406
Title: An Open-label, Multicenter Phase II Clinical Study to Evaluate Safety, Efficacy and PK of HLX208 (BRAF V600E Inhibitor) in Advanced Solid Tumor With BRAF V600 Mutation
Brief Title: A Phase II Clinical Trial to Evaluate HLX208 in Advanced Solid Tumor Patients With BRAF V600 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-ST201
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 (Experimental)
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — 900mg bid po

SUMMARY:
An Open-label, Multicenter Phase II Clinical Study to Evaluate Safety, Efficacy and PK of HLX208 (BRAF V600E Inhibitor) in Advanced Solid Tumor With BRAF V600 Mutation

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y
* Good Organ Function
* Expected survival time ≥ 3 months
* advanced solid tumors with BRAF V600 mutation that have been diagnosed
* Previous failure to standard treatment, absence of standard treatment, or insuitability for standard treatment at this stage.
* ECOG score 0-1;

Exclusion Criteria:

* Previous treatment with BRAF inhibitors or MEK inhibitors
* Symptomatic brain or meningeal metastases (unless the patient has beenon > treatment for 6 months, has no evidence of progress on imagingwithin 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable)
* A history of other malignancies within two years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin
* Patient with non-small cell lung cancer, anaplastic thyroid cancer, malignant primary intracranial tumor, melanoma, colorectal cancer or hematological tumor（Vulva and vaginal melanoma are excluded.）
* Severe active infections requiring systemic anti-infective therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | from first dose to the last patient was followed up for 6 month
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the e RECIST Version 1.1)

SECONDARY OUTCOMES:
PFS | [Time Frame: from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier)，assessed up to 1 years]
  Progression-free survival(PFS):assessed by IRRC and the investigator based on the RECIST Version 1.1
DOR | [Time Frame: from the first occurrence of a documented CR or PR (whichever recorded earlier) to the time of first documented disease progression or death (whichever occurs first) assessed up to 1 years]
  Duration of response
OS | [Time Frame: from the first dose to the time of death due to any cause，assessed up to 2 years]
  Overall survival